CLINICAL TRIAL: NCT05472090
Title: A Phase 2, 14-week Double-Blind, Randomized, Multicenter, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TNX-102 SL Taken Daily at Bedtime in Patients With Multisite Pain Associated With Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: A Phase 2 Study to Evaluate the Efficacy and Safety of TNX-102 SL in Patients With Multi-Site Pain Associated With Post-Acute Sequelae of SARS-CoV-2 Infection
Acronym: PREVAIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-CY-PA201
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Post-Acute Sequelae of SARS-CoV-2 (PASC) Infection; COVID-19; Long COVID; Long Haul COVID
Keywords: Multi-site pain; Sleep disturbance; PASC; COVID-19; Long COVID; Coronavirus infections
MeSH Terms: conditions — Infections; COVID-19; Post-Acute COVID-19 Syndrome; Parasomnias; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNX-102 SL Tablet, 5.6 mg (Experimental): 1 x TNX-102 SL 2.8 mg Tablet taken sublingually each day at bedtime for 2 weeks, then 2 x TNX-102 SL 2.8 mg (5.6 mg) Tablet taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: TNX-102 SL
- Placebo SL Tablet (Placebo Comparator): 1 x Placebo Tablet taken sublingually each day at bedtime for 2 weeks, then 2 x Placebo Tablet taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: Placebo SL Tablet

INTERVENTIONS:
Drug: TNX-102 SL — Patients will take 1 tablet of randomly assigned study drug sublingually starting on Day 1 for 2 weeks. At the Week 2 visit, all patients will have the dose increased to 2 tablets for 12 weeks.
  Arms: TNX-102 SL Tablet, 5.6 mg
Drug: Placebo SL Tablet — Patients will take 1 tablet of randomly assigned study drug sublingually starting on Day 1 for 2 weeks. At the Week 2 visit, all patients will have the dose increased to 2 tablets for 12 weeks.
  Arms: Placebo SL Tablet

SUMMARY:
This is a Phase 2, randomized, parallel-group, double-blind, placebo-controlled, 14-week study designed to evaluate the efficacy and safety of TNX-102 SL 5.6 mg (2 x 2.8 mg tablets) taken once daily at bedtime for the management of multi-site pain associated with Long COVID.

ELIGIBILITY:
Major Inclusion Criteria:

* The patient is male or female, 18 to 65 years of age, inclusive.
* The patient has a polymerase chain reaction (PCR) confirmed history of SARS-CoV-2 infection at least 3 months prior to enrollment, based on a documented written positive viral test at the time of active infection.
* The patient has new onset or significant worsening of pain that coincides with a prior COVID-19 infection and has symptoms that have been generally present for at least 3 months but no longer than 18 months.

Major Exclusion Criteria:

* The patient has been diagnosed with infectious or inflammatory arthritis (eg, rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis), systemic lupus erythematosus, untreated or active gout (ie, any acute attack within past 2 years is exclusionary), or meets criteria for another type of systemic autoimmune disease (eg, Sjogren's disease).
* The patient has been diagnosed with a complex regional pain syndrome, fibromyalgia, failed back surgery syndrome, persistent or prevalent pain symptoms related to systemic disease (eg, diabetic peripheral neuropathy, post-herpetic neuropathy), untreated hyperparathyroidism, or a history of prior surgery, trauma, organ or tissue damage, or other source of pain that, in the Investigator's opinion, would confound or interfere with the assessment of the patient's symptoms or require excluded therapies during the patient's study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herb Harris, MD, PhD, Study Director — Tonix Pharmaceuticals
Locations (28):
- United States (28):
  - Accel Research-Birmingham Clinical Research Unit, Birmingham, Alabama
  - Tonix Clinical Site, Oceanside, California
  - Tonix Clinical Site, Santa Ana, California
  - Tonix Clinical Site, Centennial, Colorado
  - Tonix Clinical Site, Aventura, Florida
  - Tonix Clinical Site, Fort Myers, Florida
  - Tonix Clinical Site, Orlando, Florida
  - Tonix Clinical Site, St. Petersburg, Florida
  - Tonix Clinical Site, Alpharetta, Georgia
  - Tonix Clinical Site, Atlanta, Georgia
  - Tonix Clinical Site, Chicago, Illinois
  - Tonix Clinical Site, Des Moines, Iowa
  - Tonix Clinical Site, Iowa City, Iowa
  - Tonix Clinical Site, Prairie Village, Kansas
  - Tonix Clinical Site, New Orleans, Louisiana
  - Tonix Clinical Site, Prairieville, Louisiana
  - Tonix Clinical Site, Boston, Massachusetts
  - Tonix Clinical Site, Methuen, Massachusetts
  - Tonix Clinical Site, Gulfport, Mississippi
  - Tonix Clinical Site, Albuquerque, New Mexico
  - Tonix Clinical Site, New York, New York
  - Tonix Clinical Site, Williamsville, New York
  - Tonix Clinical Site, Shelby, North Carolina
  - Tonix Clinical Site, Columbus, Ohio
  - Tonix Clinical Site, Dayton, Ohio
  - Tonix Clinical Site, Tulsa, Oklahoma
  - Tonix Clinical Site, Austin, Texas
  - Tonix Clinical Site, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Started | 32 | 31
Completed | 26 | 25
Not Completed | 6 | 6
Not completed — Adverse Event | 2 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (8.80) | 51.4 (10.01) | 50.0 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 11 | 6 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 21 | 24 | 45
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.78 (4.067) | 29.49 (4.439) | 29.64 (4.222)

OUTCOME MEASURES:

1. Primary Outcome: Daily Diary Pain NRS
Description: Change from Baseline in the diary Numeric Rating Scale (NRS) weekly average of daily self-reported worst Long COVID pain intensity scores at the Week 14 endpoint. Scores range from 0 to 10 where a higher score means worse outcome.
Time Frame: Week 14
Population: Intention-to-treat (ITT) population defined as all patients who were randomized and had at least one post-baseline daily diary entry.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 32 | 31
units on a scale | -2.2 (0.34) | -2.0 (0.35)

2. Secondary Outcome: Daily Diary Sleep Quality NRS
Description: Mean change from baseline in the weekly average of the daily diary numeric rating scale (NRS) assessment of sleep quality at the Week 14 endpoint. Scores range from 0 to 10 where a higher score means worse outcome.
Time Frame: Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 32 | 31
units on a scale | -2.1 (0.38) | -1.6 (0.39)

3. Secondary Outcome: PROMIS Fatigue -Short Form 8a
Description: Change from Baseline in the Patient Reported Outcomes Measurement Information System (PROMIS) score for fatigue at the Week 14 endpoint. Subjects are asked to reflect on their fatigue symptoms in the past 7 days and respond to 8 questions on a 5 point scale (1 to 5) where a higher score indicates a worse outcome. The total score is reported on a range of 8 to 40. Raw scores are converted to T-scores based on US population with score of 50 as average with a standard deviation of 10.
Time Frame: Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 32 | 31
T-score | -8.0 (1.65) | -3.2 (1.68)

4. Secondary Outcome: PROMIS Cognitive Function - Abilities-Short Form 8a
Description: Change from Baseline in the Patient Reported Outcomes Measurement Information System (PROMIS) score for cognitive function at the Week 14 endpoint. Subjects are asked to reflect on their cognitive function and abilities in the past 7 days and respond to 8 questions on a 5 point scale (1 to 5) where a higher score indicates a worse outcome. The total score is reported on a range of 8 to 40. Raw scores are converted to T-scores based on US population with score of 50 as average with a standard deviation of 10.
Time Frame: Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 32 | 31
T-score | 5.4 (1.55) | 3.5 (1.55)

ADVERSE EVENTS:
Time Frame: Patients were monitored for AEs throughout the study. The total duration of the study, including screening and follow up, was as long as 25 weeks.
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 12/32 | 2/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TNX-102 SL Tablet, 5.6 mg (N=32) | Placebo SL Tablet (N=31)
Hypoaesthesia oral (Gastrointestinal disorders) | 6 | 0 — Tongue numbness
Glossodynia (Gastrointestinal disorders) | 2 | 0 — burning tongue/sensation of the tongue, tongue discomfort
Oral Pain (Gastrointestinal disorders) | 2 | 0
Paraesthesia oral (Gastrointestinal disorders) | 2 | 0
Influenza like illness (General disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
We consider the study completed and not terminated because although participant enrollment stopped early, those that were already enrolled in the study were allowed to complete treatment and all assessments and visits per protocol. Therefore, we consider that participant's last visit has occurred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all study investigators.

DOCUMENTS (2):
  • Study Protocol (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT05472090/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT05472090/SAP_001.pdf